CLINICAL TRIAL: NCT07106658
Title: Transcutaneous Electrical Acupoint Stimulation (TEAS) in Cirrhotic Patients Undergoing Urgent Endoscopy for Acute Esophagogastric Variceal Bleeding: A Randomized Controlled Trial
Brief Title: TEAS in Liver Patients Needing Urgent Endoscopy for Bleeding Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Liu Yan, Chief of Gastroenterology and Hepatology, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 302-2025-002
Record Dates: First submitted 2025-07-08; First posted 2025-08-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Endoscopy; Upper Gastrointestinal Hemorrhage
Keywords: Variceal Bleeding; Transcutaneous Electrical Acupoint Stimulation; Cirrhotic
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real TEAS + Urgent Endoscopy (Experimental): Participants receive real Transcutaneous Electrical Acupoint Stimulation (TEAS) delivered via surface electrodes bilaterally at four predefined acupoints (Hegu [LI4], Neiguan [PC6], Zusanli [ST36], Gongsun [SP4]). Stimulation (dense-disperse wave, 2/100Hz frequency, intensity 5-15mA based on tolerance) begins 30 minutes before urgent endoscopy and continues throughout the procedure. All participants receive standard medical management and urgent endoscopy.
  Interventions: Other: TEAS + Urgent Endoscopy
- Sham TEAS + Urgent Endoscopy (Sham Comparator): Participants receive placebo TEAS. Electrodes are placed identically to the Active TEAS Group at the same four acupoints (Hegu [LI4], Neiguan [PC6], Zusanli [ST36], Gongsun [SP4]) using the same device, but no electrical current is delivered. The device appears active to maintain blinding. All participants receive standard medical management and urgent endoscopy.
  Interventions: Other: Sham TEAS + Urgent Endoscopy
- Urgent Endoscopy Only (Other): Participants receive standard urgent endoscopy care only, with no TEAS electrodes or device applied. They receive identical standard medical management and urgent endoscopy as the other groups.
  Interventions: Other: Urgent Endoscopy Only

INTERVENTIONS:
Other: TEAS + Urgent Endoscopy — Participants receive real Transcutaneous Electrical Acupoint Stimulation (TEAS) delivered via surface electrodes bilaterally at four predefined acupoints (Hegu [LI4], Neiguan [PC6], Zusanli [ST36], Gongsun [SP4]). Stimulation (dense-disperse wave, 2/100Hz frequency, intensity 5-15mA based on tolerance) begins 30 minutes before urgent endoscopy and continues throughout the procedure. All participants receive standard medical management and urgent endoscopy.
  Arms: Real TEAS + Urgent Endoscopy
Other: Sham TEAS + Urgent Endoscopy — Participants receive placebo TEAS. Electrodes are placed identically to the Active TEAS Group at the same four acupoints (Hegu [LI4], Neiguan [PC6], Zusanli [ST36], Gongsun [SP4]) using the same device, but no electrical current is delivered. The device appears active to maintain blinding. All participants receive standard medical management and urgent endoscopy.
  Arms: Sham TEAS + Urgent Endoscopy
Other: Urgent Endoscopy Only — Participants receive standard urgent endoscopy care only, with no TEAS electrodes or device applied. They receive identical standard medical management and urgent endoscopy as the other groups.
  Arms: Urgent Endoscopy Only

SUMMARY:
The goal of this clinical trial is to learn if a non-invasive electrical therapy (called TEAS) applied to specific points on the skin can help patients with severe liver disease better tolerate emergency stomach scope for serious bleeding. It will also test whether TEAS improves procedural efficiency, hemostasis outcomes, and patient tolerance.

The main questions the study aims to answer are:

1. Does TEAS shorten procedure time for diagnostic and therapeutic endoscopy?
2. Does TEAS improve immediate hemostasis success and reduce early rebleeding?
3. Does TEAS reduce patient discomfort and improve procedural tolerance during urgent endoscopy?

Researchers will compare three approaches:

1. Active TEAS: Electrical stimulation at specific points on hands/legs before and during the scope..
2. Sham TEAS: Pads placed on the skin but no electrical stimulation.
3. Control: Standard procedure without any pads or stimulation.

Participants with acute upper digestive bleeding due to liver disease who need an emergency scope will:

1. Be randomly assigned to one of the three groups.
2. Receive either Real TEAS, Sham TEAS, or No TEAS just before and during their emergency stomach scope procedure.
3. Have procedural efficiency (time) and hemostasis outcomes recorded.
4. Have discomfort levels assessed using a Visual Analogue Scale (VAS).
5. Have physiological parameters (heart rate, blood pressure, respiratory rate) monitored.
6. Be evaluated for endoscopic success, patient satisfaction, and clinical experience measures.

Researchers will watch for any side effects from the TEAS pads or the procedure.

DETAILED DESCRIPTION:
Background and Rationale:

Acute esophagogastric variceal bleeding (AEGVB) in cirrhotic patients is a life-threatening emergency requiring urgent endoscopic intervention. Emergency endoscopy, often performed under conscious sedation or minimal anesthesia due to the urgency and patient instability, is associated with significant patient discomfort, poor tolerance, hemodynamic fluctuations (tachycardia, hypertension), nausea/vomiting, and compromised procedural success. This discomfort can lead to suboptimal visualization, incomplete treatment, and increased risk of complications. Effective, low-risk adjunctive methods to improve tolerance and stability during this critical procedure are needed. Transcutaneous Electrical Acupoint Stimulation (TEAS) is a non-invasive modality derived from traditional acupuncture principles, delivering controlled electrical currents to specific acupoints via surface electrodes. Preliminary evidence suggests TEAS may reduce procedural discomfort, promote hemodynamic stability, regulate gastrointestinal function, and potentially enhance hemostasis. However, robust evidence on its efficacy and safety specifically during urgent endoscopy for AEGVB in cirrhotic patients is lacking. This trial aims to rigorously evaluate whether adjunctive TEAS improves procedural tolerance and clinical outcomes in this high-risk population.

Study Design and Methodology:

This is a prospective, randomized, single-center, three-arm, controlled trial. Cirrhotic patients presenting with EGVB requiring urgent endoscopy within 48 hours will be assessed for eligibility. Eligible and consenting participants will be randomly assigned (1:1:1) using computer-generated random numbers with allocation concealment to one of three groups:

Active TEAS Group: Receives real TEAS stimulation applied bilaterally to four predefined acupoints (Hegu [LI4], Neiguan [PC6], Zusanli [ST36], Gongsun [SP4]) using a standardized device (dense-disperse wave, 2/100Hz frequency, intensity adjusted to patient tolerance [typically 5-15mA]). Stimulation begins 10 minutes before endoscope insertion and continues throughout the endoscopic procedure.

Sham TEAS Group: Receives identical electrode placement at the same acupoints using the same device, but no electrical current is delivered (device appears active). This controls for the placebo effect of device application and acupressure.

Control Group: Receives standard urgent endoscopy care without any TEAS electrodes or device application.

All participants receive standardized pre-endoscopic medical management (fluid resuscitation, vasoactive drugs, antibiotics as indicated) and undergo the urgent endoscopic procedure (diagnostic and therapeutic) performed by experienced endoscopists blinded to group assignment, using institutional protocols. The TEAS/sham operator is not involved in outcome assessment.

Primary Focus:

The study primarily investigates whether active TEAS, compared to sham or standard care:

1. Enhances procedural efficiency: Measured as total endoscopy time for diagnostic and therapeutic procedures.
2. Improves hemostasis outcomes: Including immediate hemostasis success and 7-day rebleeding rate.
3. Ameliorates procedural tolerance: Assessed via patient-reported discomfort (VAS), endoscopy success rate, and physiological stability.

Safety Monitoring:

Adverse events related to TEAS (e.g., local skin irritation, pain at electrode sites) and the endoscopic procedure (e.g., aspiration, perforation) are meticulously recorded and managed per protocol.

Scientific Justification:

The selection of specific acupoints (LI4, PC6, ST36, SP4) is based on traditional Chinese medicine principles and modern physiological understanding: targeting points associated with analgesia (LI4, PC6), gastrointestinal motility regulation and anti-emesis (PC6, ST36), hemodynamic stabilization (PC6), and potential enhancement of hemostatic mechanisms (SP4, ST36). The sham-controlled design is crucial for isolating the specific effects of electrical neuromodulation from non-specific placebo effects. This trial addresses a significant gap in optimizing the high-stakes scenario of urgent endoscopy for AEGVB by evaluating a readily deployable, non-pharmacological adjunctive strategy.

ELIGIBILITY:
1. Inclusion Criteria:

1. Patients aged 18-80 years with suspected or confirmed esophageal-gastric variceal bleeding (EGVB);
2. Patients with confirmed cirrhosis (any etiology/Child-Pugh class) presenting with upper gastrointestinal hemorrhage.

2. Exclusion Criteria:

1. Neuropsychiatric disorders preventing valid assessment:

   Hepatic encephalopathy ≥Grade II Severe anxiety Cognitive impairment
2. High-risk physiological status:

   ASA class >III Hemodynamic instability (systolic BP <90 mm Hg after resuscitation)
3. Contraindications for TEAS/emergency care:

   Skin lesions at acupoints Electrical implants Allergies to TEAS electrodes/emergency medications
4. Pregnant or lactating women;
5. History of long-term alcohol/opioid abuse;
6. Inability to provide informed consent;
7. Prior TEAS experience (to maintain blinding integrity).

3. Dropout Criteria:

1. Serious TEAS/endoscopy-related adverse reactions:

   Severe allergic reactions Hemodynamic collapse
2. Life-threatening deterioration during endoscopy:

   Uncontrolled bleeding Respiratory failure Hepatic encephalopathy progression
3. Principal investigator-identified safety risks (e.g., sepsis, acute liver failure);
4. Inability to complete protocols due to emergent complications:

   Intubation Altered mental status ICU transfer
5. Voluntary withdrawal by participant/legal representative.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Procedural Efficiency | Immediately after the endoscopy procedure
  Total endoscopy time (minutes), recorded from scope insertion to withdrawal, analyzed separately for diagnostic-only procedures and therapeutic interventions.
Hemostasis Outcomes | Within 7 days post-procedure
  1. Immediate hemostasis success: Defined as cessation of active bleeding observed at procedure completion.
  2. 7-day rebleeding rate: Defined as clinically significant bleeding from the same source within 7 days post-procedure.

SECONDARY OUTCOMES:
Discomfort Level | At 30 minutes post-procedure
  A self-made questionnaire comprising five visual analogue scales (VASs) evaluated discomfort across nausea and vomiting, throat discomfort, bucking, abdominal distension/pain, and agitation. Each VAS was a 10 cm horizontal line segment scored from 0 (no discomfort) to 10 (highest discomfort intensity), where patients marked their perceived level for each symptom. All participants completed the five VASs at 30 minutes post-procedure, and the mean score was calculated.
Blood pressure | At pre-endoscopy (baseline), during active endoscopy, and 30 minutes post-procedure
  Blood pressure is measured in millimeters of mercury (mmHg). Systolic blood pressure and diastolic blood pressure were continuously monitored also using a multiparameter patient monitor (Type Prince-100B, Heal Force Bio-meditech Holdings Limited, China). Measurements were recorded at three phases: pre-endoscopy (baseline), during active endoscopy, and 30 minutes post-procedure to evaluate hemodynamic responses to the intervention.
Heart rate | At pre-endoscopy (baseline), during active endoscopy, and 30 minutes post-procedure
  Heart rate (unit of measure: beat per minute) was continuously monitored using a multiparameter patient monitor (Type Prince-100B, Heal Force Bio-meditech Holdings Limited, China). Measurements were recorded at three phases: pre-endoscopy (baseline), during active endoscopy, and 30 minutes post-procedure to evaluate hemodynamic responses to the intervention.
Procedural Tolerance | Immediately after the endoscopy procedure
  A composite endpoint of endoscopy success, requiring both technical adequacy (complete visualization score 4/4) and patient satisfaction (Likert score ≤ 2).

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Lu, Doctor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
1. Ongoing Research Commitments Further analyses and secondary studies using the same dataset are planned, including subgroup investigations and long-term outcome assessments. Premature data sharing could compromise the integrity of these planned works.
  2. Participant Privacy and Confidentiality The dataset contains sensitive clinical information (e.g., cirrhosis etiology, hemorrhage severity, neuropsychiatric status). Complete anonymization is challenging, and re-identification risks violate ethical/legal safeguards.

REFERENCES:
- [Background] Cheong YC, Dix S, Hung Yu Ng E, Ledger WL, Farquhar C. Acupuncture and assisted reproductive technology. Cochrane Database Syst Rev. 2013 Jul 26;2013(7):CD006920. doi: 10.1002/14651858.CD006920.pub3. PMID 23888428
- [Background] Lee H, Ernst E. Acupuncture for GI endoscopy: a systematic review. Gastrointest Endosc. 2004 Nov;60(5):784-9. doi: 10.1016/s0016-5107(04)02030-9. No abstract available. PMID 15557955